CLINICAL TRIAL: NCT02505269
Title: Brentuximab Vedotin Plus AD in Non-bulky Limited Stage Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Seagen Inc. (Industry)
Responsible Party: Principal Investigator, Jeremy Abramson, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-196
Record Dates: First submitted 2015-07-20; First posted 2015-07-22 (Estimated); Results first posted 2020-08-24 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Hodgkin Lymphoma
Keywords: limited stage; Hodgkin's disease; non-bulky
MeSH Terms: conditions — Hodgkin Disease | interventions — Brentuximab Vedotin; Doxorubicin; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Brentuximab Vedotin (Experimental): The following procedures will take place during study visits beginning after the screening procedures:
  - Participants will receive combination therapy:
  * Brentuximab Vedotin intravenously on predetermined days per cycle
  * Adriamycin intravenously on predetermined days per cycle
  * Dacarbazine intravenously on predetermined days per cycle
  Interventions: Drug: Brentuximab Vedotin; Drug: Adriamycin; Drug: Dacarbazine

INTERVENTIONS:
Drug: Brentuximab Vedotin
  Other Names: Adcetris
Drug: Adriamycin
  Other Names: Doxorubicin; Rubex ®
Drug: Dacarbazine
  Other Names: DTIC-Dome®; DTIC; DIC; Imidazole Carboxamide

SUMMARY:
Limited stage Hodgkin lymphoma is a highly curable disease, but standard treatment with ABVD chemotherapy and radiation can lead to late risks of secondary cancers, lung injury, heart injury, and others. This trial eliminates radiation therapy and reduces intensity of chemotherapy by incorporating the highly active FDA-approved targeted therapy brentuximab vedotin, an antibody-drug conjugate specifically against the lymphoma cells, combined with the standard chemotherapy drugs Adriamycin and Dacarbazine (AD).

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied. It also means that the FDA (the U.S. Food and Drug Administration) has not yet approved brentuximab vedotin (brentuximab) as part of the initial treatment of Hodgkin lymphoma. Currently, brentuximab is FDA-approved for treatment of relapsed Hodgkin lymphoma.

* Brentuximab works by binding specifically to Hodgkin lymphoma cells, entering the cells, and then releasing the drug to destroy the cell.
* The chemotherapy drugs Adriamycin and Dacarbazine (AD) which which participants will receive in this research study are approved for use in people with Hodgkin Lymphoma.
* Patients will not receive planned radiation therapy, or the drugs bleomycin or vinblastine.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated stage IA, IB, or IIA classical Hodgkin Lymphoma
* Non-bulky disease defined as less than 10 cm in maximal diameter
* Measurable disease ≥1.5 cm
* Age ≥18
* ECOG performance status 0-2 (see Appendix B)
* Participants must have initial organ and marrow function as defined below:

  * Absolute neutrophil count ≥ 1,000/mcL
  * Platelets ≥100,000/mcL
  * Total bilirubin ≤ 2, unless due to Gilbert's disease
  * AST (SGOT)/ALT (SGPT) ≤ 2.5 X institutional upper limit of normal
  * Creatinine clearance ≥ 30 mL/min
* LVEF by echocardiogram or MUGA within institutional normal limits
* Participant must be willing to use two effective forms of birth control during protocol therapy. Men and women must continue using two effective forms of birth control for 6 months following treatment.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Participants who have had prior cHL-directed chemotherapy or radiotherapy
* Participants may not be receiving any other investigational agents
* Participants with known CNS involvement of lymphoma
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Adriamycin, Dacarbazine, or brentuximab
* Pre-existing grade 2 or greater neuropathy
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because brentuximab is an antibody drug conjugate with a linked potent anti-tubule agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother with brentuximab, breastfeeding should be discontinued if the mother is treated with brentuximab. These potential risks may also apply to other agents used in this study.
* Participants with a history of a different malignancy are ineligible unless they have been disease free for 1 year and considered at low risk for relapse, except for: cervical cancer in situ, ductal carcinoma in situ, localized prostate cancer with no detectable disease by imaging studies, and non-melanoma cancers of the skin, which are eligible at any time.
* Known HIV positivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-08-07 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Abramson, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Derived] Abramson JS, Bengston E, Redd R, Barnes JA, Takvorian T, Sokol L, Lansigan F, Armand P, Shah B, Jacobsen E, Martignetti R, Turba E, Metzler S, Patterson V, LaCasce AS, Bello CM. Brentuximab vedotin plus doxorubicin and dacarbazine in nonbulky limited-stage classical Hodgkin lymphoma. Blood Adv. 2023 Apr 11;7(7):1130-1136. doi: 10.1182/bloodadvances.2022008420. PMID 36053786

RESULTS

PARTICIPANT FLOW:
Groups:
- Brentuximab Vedotin: The following procedures will take place during study visits beginning after the screening procedures:
  - Participants will receive combination therapy:
  * Brentuximab Vedotin intravenously on predetermined days per cycle
  * Adriamycin intravenously on predetermined days per cycle
  * Dacarbazine intravenously on predetermined days per cycle
  Brentuximab Vedotin
  Adriamycin
  Dacarbazine
Period: Overall Study
Arm/Group | Brentuximab Vedotin
Started | 34
Completed | 34
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 34
Age, Continuous [Median (Full Range); unit: years] | 36 [18 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate
Description: The number of patients that achieved a complete response (CR) to therapy as assessed by the revised International Working Group Criteria.
  Complete response:
  * Lymph nodes and extralymphatic sites: Score 1, 2, or 3 with or without a residual mass on 5-point (Daeuville) scale
  * Bone Marrow: No evidence of FDG-avi disease
  * No new lesions
  Deauville Criteria for PET scan Interpretation in Lymphoma
  Five-point scale:
  1. No Uptake
  2. Uptake ≤ mediastinum
  3. Uptake >mediastinum but ≤ liver
  4. Uptake moderately increased compared to liver at any site
  5. Uptake markedly increased compared to the liver at any site or/and new sites of disease
Time Frame: 4-6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 34
Participants | 34

2. Secondary Outcome: Overall Response Rate
Description: The number of patients that achieved a complete Metabolic Response (CR) or Partial Metabolic Response (PR) to therapy as assessed by the revised International Working Group Criteria.
  Complete Metabolic Response:
  Lymph nodes and extralymphatic sites: Score 1, 2, or 3 with or without a residual mass on 5-point (Daeuville) scale Bone Marrow: No evidence of FDG-avi disease No new lesions
  Partial Metabolic Response:
  >Lymph nodes and extralymphatic sites: Score 4, 5 with reduced uptake compared with baseline and residual mass(es) of any size.
  Deauville Criteria for PET scan Interpretation in Lymphoma
  Five-point scale:
  1. No Uptake
  2. Uptake ≤ mediastinum
  3. Uptake >mediastinum but ≤ liver
  4. Uptake moderately increased compared to liver at any site
  5. Uptake markedly increased compared to the liver at any site or/and new sites of disease
Time Frame: 4-6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 34
Participants | 34

3. Secondary Outcome: Number of Patients With Grade III and IV Adverse Events
Description: The number of patients that experienced grade III and grade IV adverse events that were deemed to be possibly, probably, or definitely related to study treatment. Adverse events were assessed using Common Toxicology Criteria for Adverse Events (CTCAE v4.0) criteria.
Time Frame: 4-6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 34
Participants
  Grade III Adverse Events | 4
  Grade IV Adverse Events | 0

ADVERSE EVENTS:
Time Frame: From the start of treatment until 30 days after the end of treatment (up to approximately 5 months)
Arm/Group | Brentuximab Vedotin
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 5/34
Other Adverse Events (participants affected / at risk) | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brentuximab Vedotin (N=34)
Colitis (Gastrointestinal disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Upper respiratory infection (Infections and infestations) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Thromboembolic event (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brentuximab Vedotin (N=34)
Abdominal pain (Gastrointestinal disorders) | 5 (6)
Alanine aminotransferase increased (Investigations) | 7 (9)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 12 (14)
Anemia (Blood and lymphatic system disorders) | 5 (6)
Anorexia (Metabolism and nutrition disorders) | 6 (7)
Anxiety (Psychiatric disorders) | 9 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (7)
Aspartate aminotransferase increased (Investigations) | 7 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Bloating (Gastrointestinal disorders) | 2 (4)
Blurred vision (Eye disorders) | 2 (2)
Breast pain (Reproductive system and breast disorders) | 2 (2)
Concentration impairment (Nervous system disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 18 (24)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Dry eye (Eye disorders) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3)
Dysgeusia (Nervous system disorders) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 6 (9)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (7)
Endocrine disorders - Other, specify (Endocrine disorders) | 3 (3)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 (2)
Fatigue (General disorders) | 21 (29)
Fever (General disorders) | 3 (3)
Flushing (Vascular disorders) | 3 (4)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 5 (6)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 5 (5)
General disorders and administration site conditions - Other, specify (General disorders) | 2 (3)
Gingival pain (Gastrointestinal disorders) | 2 (3)
Headache (Nervous system disorders) | 9 (13)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hot flashes (Vascular disorders) | 4 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (7)
Insomnia (Psychiatric disorders) | 2 (2)
Lymphocyte count decreased (Investigations) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 6 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Nausea (Gastrointestinal disorders) | 27 (39)
Neck edema (General disorders) | 2 (4)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Neutrophil count decreased (Investigations) | 8 (11)
Non-cardiac chest pain (General disorders) | 4 (5)
Paresthesia (Nervous system disorders) | 5 (6)
Peripheral sensory neuropathy (Nervous system disorders) | 21 (29)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (8)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8 (16)
Scalp pain (Skin and subcutaneous tissue disorders) | 3 (3)
Skin ulceration (Skin and subcutaneous tissue disorders) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Tinnitus (Ear and labyrinth disorders) | 2 (2)
Upper respiratory infection (Infections and infestations) | 4 (4)
Vomiting (Gastrointestinal disorders) | 5 (5)
White blood cell decreased (Investigations) | 6 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-23): https://cdn.clinicaltrials.gov/large-docs/69/NCT02505269/Prot_SAP_000.pdf